CLINICAL TRIAL: NCT02406456
Title: Real-time fMRI Neurofeedback as a Treatment Tool for Alcohol Dependence - Protocol Optimisation Phase
Brief Title: Optimisation of Functional MRI-based Neurofeedback for Alcohol Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff University (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, David Linden, Professor of Translational Neuroscience, Cardiff University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRAINTRAINPILOT
Record Dates: First submitted 2015-03-26; First posted 2015-04-02 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Alcohol Abuse
MeSH Terms: conditions — Alcoholism | interventions — Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neurofeedback (Experimental)
  Interventions: Other: Neurofeedback

INTERVENTIONS:
Other: Neurofeedback

SUMMARY:
Participants will undergo a single session of functional magnetic resonance imaging (fMRI)-based neurofeedback (approximately 1 hour). The investigators will assess their ability to regulate motivational networks of the brain during the exposure to alcohol cues and evaluate immediate effects on craving and cognitive bias for alcohol by administering a questionnaire and a Stroop task before and after the session.

ELIGIBILITY:
Inclusion Criteria:

* History of alcohol use disorder or current alcohol consumption above 21 units (1 unit = 8g) of alcohol per week (male participants) or above 14 units of alcohol per week (female participants)

Exclusion Criteria:

* MRI safety exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Neurofeedback success (brain activation difference during neurofeedback and baseline blocks) | 1 day
  This measure will be based on the analysis of participants' fMRI (functional magnetic resonance imaging) data, reflecting brain activation, during exposure to alcohol cues. Neurofeedback success will be defined as significant difference between activation levels (expressed as beta weights of a linear regression model) during the regulation periods compared to baseline. The significance will be determined by a t-test.

SECONDARY OUTCOMES:
Drinking Urges Questionnaire as a measure of alcohol craving | 1 day
  Measure of alcohol craving
Alcohol Stroop task as a measure of cognitive bias | 1 day
  Measure of cognitive bias

CONTACTS AND LOCATIONS:
Overall Officials: David Linden, MD, Principal Investigator — Cardiff University
Locations (1):
- School of Medicine, Cardiff University, Cardiff, Wales, United Kingdom